CLINICAL TRIAL: NCT00448747
Title: A Multi-center, Study Investigating a New, Oral Growth Hormone Secretagogue (GHS)(AEZS 130, Formerly Ardana (ARD)-07) as a Growth Hormone (GH) Stimulation Test in Terms of Safety and Efficacy
Brief Title: Investigation of a New, Oral Growth Hormone Secretagogue, AEZS-130 as a Growth Hormone Stimulation Test.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: AEZS 130 047
Record Dates: First submitted 2007-03-16; First posted 2007-03-19 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2017-06

CONDITIONS: Diagnosis of Adult Growth Hormone Deficiency (AGDH)
Keywords: Ghrelin mimetic, growth hormone secretagogue
MeSH Terms: interventions — macimorelin

STUDY DESIGN:
Intervention Model Description: Multi-center, randomized, open-label, cross-over trial to compare AEZS-130 to an established GH stimulation test, L-ARG+GHRH, in the diagnosis of GH deficiency and in terms of safety. Following Amendment no. 3 (version 27 May 2010) , no cross-over was performed anymore due to unavailability of L-ARG+GHRH with resulting single arm testing of AEZS-130. Thus, two treatment arms were applicable only as long as GHRH as substance was available.
Oversight: Data Monitoring Committee: No

ARMS (2):
- AEZS-130 ( formerly ARD-07) (Experimental): A single oral administration of AEZS-130 (0.5 mg/kg po) as Growth Hormone Stimulation Test
  Interventions: Drug: AEZS-130 (formerly ARD-07)
- L-ARG+GHRH (Active Comparator): This trial was set up as a multi-center, randomized, cross-over study investigating AEZS-130 as a Growth Hormone Stimulation Tests in terms of safety and efficacy compared to L-ARG+GHRH. When GHRH became unavailable on the US market, this comparator arm was no longer available, which was addressed by Amendment No. 3 (version 27-March-2010). Control subject enrolled under Amendment No. 3 were not randomized as there was no cross-over due to unavailability of L-ARG+GHRH. These control subjects received only AEZS-130
  Interventions: Drug: L-ARG+GHRH

INTERVENTIONS:
Drug: AEZS-130 (formerly ARD-07) — A single oral administration of AEZS-130 as Growth Hormone Stimulation Test
  Other Names: Test 1; Macimorelin
  Arms: AEZS-130 ( formerly ARD-07)
Drug: L-ARG+GHRH — A single administration of L-ARG+GHRH (iv bolus) followed by a 30min infusion of L-ARG as Growth Hormone Stimulation Test
  Other Names: Test Control
  Arms: L-ARG+GHRH

SUMMARY:
The diagnosis of growth hormone deficiency (GHD) in adults is established by laboratory testing in patients with an appropriate clinical history of hypothalamic pituitary disease. Two tests that are considered to be gold standard tests for the diagnosis of GHD are the insulin tolerance test (ITT) and growth hormone releasing hormone (GHRH) combined with L-arginine (L-ARG). However, these tests are either bothersome (given intravenously) to the patient or are linked with side effects. Therefore, an orally available compound like AEZS-130 (formerly ARD-07), if demonstrated to be safe and providing adequate sensitivity and specificity could be a welcome alternative and/or complement to the current available tests.

The intent was to recruit 40 adult GHD (AGHD) patients and 40 healthy control subjects into this trial, but the original sponsor (Ardana Biosciences Ltd.) discontinued the study for financial reasons before this was completed. At the time of withdrawal of GHRH from the market in 2008, 42 AGHD patients and 10 normal controls had completed the study at 9 US sites. This study reactivated to complete the remaining 30 matched control subjects.

Additionally upon agreement with the FDA in a Special Protocol Assessment (SPA), 10 additional adult growth hormone deficient and their matched control were planned to be enrolled into this trial for a total treated population of approximatively 100 subjects.

DETAILED DESCRIPTION:
Thirty control subjects (i.e., without AGHD) were matched to the 30 AGHD patients who were not previously matched. Matching was based upon gender, age, BMI, and estrogen status for females. They received one oral dose of AEZS-130 followed by serial blood draws for growth hormone (GH), insulin-like growth factor 1 (IGF-1) and pharmacokinetic (PK) determinations. There was no cross over due to the unavailability of GHRH (Geref) in the United States. Under Amendment #4 to this protocol, 10 additional AGHD subjects were to be enrolled and matched as described above.

Furthermore, the objective of the study was changed to delete comparison with L-ARG + GHRH.

ELIGIBILITY:
Inclusion for Matched Control Subjects:

* Undergone normal growth and development
* Normal serum prolactin (PRL) concentrations
* Females should have a history of regular, age-appropriate menses
* Males should have normal serum testosterone concentrations
* Matched GHD subject already enrolled in study; matched in terms of sex, age, BMI and Estrogen status (women only)

Exclusion Criteria for Matched Control Subjects:

* Inability or unwillingness to comply with study medication
* Pregnancy or lactation
* Clinically relevant ECG abnormalities (including QT/QTc interval > 450 ms) at any time prior to dosing at Visit 2
* Treatment with any drugs that might prolong QT/QTc

Inclusion criteria dor Adult GHD Subjects:

* Confirmed GH deficiency with a low IGF-1
* 3 months of stable treatment for those requiring hormone replacement therapy for hormones deficiencies other than GHD
* subjects with hypogonadism must be treated with sex steroid therapy, excluding women over 50 yr of age
* women on estrogen therapy, for whatever reason, must be on stable treatment for ar least 3 months prior to study

Exclusion criteria for Adult GHD Subjects:

* Untreated hypothyroidism
* Known hypersensitivity to any excipient in study medication
* Inability or unwillingness to comply with study procedures
* Intracranial lesions stable for less than 12 months
* GH therapy within one month of study entry
* Clinically significant cardiovascular, or cerebrovascular disease
* Current active malignancy other than non-melanoma skin cancer
* Renal or hepatic dysfunction (> 3 x ULN liver function enzymes (LFEs) - aspartate amino transferase (ASAT); alanine amino transferase (ALAT); gamma-glutamyltransferase (GGT) or creatinine > 2x ULN)
* Pregnancy or lactation
* Active Cushing's disease
* Clinically relevant ECG abnormalities (including QT/heart rate corrected QT interval (QTc) interval > 450 ms) at any time prior to dosing at Visit 2
* Treatment with any drugs that might prolong QT/QTc

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2007-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beverly MK Biller, MD, Principal Investigator — Massachusetts General Hospital, Boston
Locations (13):
- United States (13):
  - Celerion, Tempe, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Northwestern University, Chicago, Illinois
  - Radiant Research Inc., Chicago, Illinois
  - John Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Celerion, Lincoln, Nebraska
  - Celerion, Neptune City, New Jersey
  - Oregon Health & Science University, Portland, Oregon
  - Baylor College of Medicine, Houston, Texas
  - Cetero Research, San Antonio, Texas
  - VA Puget Sound HCS University of Washington, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No
To share IPD is not planned as subjects were not informed about this possibility and thus, no related patient consent is available (data protection issue).

REFERENCES:
- [Result] Garcia JM, Swerdloff R, Wang C, Kyle M, Kipnes M, Biller BM, Cook D, Yuen KC, Bonert V, Dobs A, Molitch ME, Merriam GR. Macimorelin (AEZS-130)-stimulated growth hormone (GH) test: validation of a novel oral stimulation test for the diagnosis of adult GH deficiency. J Clin Endocrinol Metab. 2013 Jun;98(6):2422-9. doi: 10.1210/jc.2013-1157. Epub 2013 Apr 4. PMID 23559086

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 53 AGHD patients and 48 matched control subjects were enrolled at 11 centers across the United States, and all subjects, with the exception of 1 AGHD patient, received macimorelin and completed the study.
  In Amendment No. 4, the objective of the study was changed to delete the comparison with L-ARG + GHRH.
Groups:
- AGHD Patients (= Cases): All Adult Growth Hormone Deficiency (AGHD) patients enrolled in the study.
- Matched Controls (= Controls): All matched control subjects enrolled in the study.
Period: Overall Study
Arm/Group | AGHD Patients (= Cases) | Matched Controls (= Controls)
Started (Safety Analysis Set: all subjects enrolled; one subject included who had not received AEZS-130.) | 53 | 48
Received First Drug Administration | 53 | 48
Received Second Drug Administration | 42 | 10
Received AEZS-130 | 52 | 48
Received L-ARG-GHRH | 43 | 10
Received L-ARG-GHRH and AEZS-130 | 42 | 10
Per Protocol Population (PPS) | 50 | 48
Completed (modified Intention-to-treat (mITT) population) | 52 | 48
Not Completed | 1 | 0
Not completed — collapsed veins | 1 | 0

BASELINE CHARACTERISTICS:
Population: Saftey Analysis Set. This is including one case (AGHD patient) who did not receive AEZS-130.
Groups:
- AGHD Patients (= Cases): All AGHD patients enrolled in the study.
- Total: Total of all reporting groups
Arm/Group | AGHD Patients (= Cases) | Matched Controls (= Controls) | Total
Number analyzed (Participants) | 53 | 48 | 101
Age, Customized [Count of Participants; unit: Participants]
  < 50 years | 27 | 19 | 46
  >= 50 years | 26 | 29 | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 61
  Male | 22 | 18 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 49 | 29 | 78
  Black or African American | 2 | 18 | 20
  Asian | 2 | 0 | 2
  Other | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53 | 48 | 101
Body Mass Index (kg/m^2) [Count of Participants; unit: Participants]
  Lean (<25) | 7 | 7 | 14
  Overweight (>=25 and <30) | 15 | 13 | 28
  Obese (>=30) | 31 | 28 | 59
Etiology of AGHD [Number; unit: participants]
  Pituitary Adenoma | 34 | 0 | 34
  CNS tumors | 8 | 0 | 8
  Others | 18 | 0 | 18

OUTCOME MEASURES:

1. Primary Outcome: Receiver Operating Characteristic (ROC) Analysis on Peak GH (Growth Hormon) Concentrations
Description: The primary endpoint for each individual is the peak GH concentration following AEZS-130 (macimorelin) administration.
Time Frame: GH sampling: pre-dose and 30, 45, 60, 75, 90, 120, 150 min post-dose
Population: PPS = per protocol set: this was considered to be the most appropriate for determination of the diagnostic utility of macimorelin
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cases/AEZS-130 Administered: All AGHD patients who were enrolled in the study and following macimorelin administration.
- Control/AEZS-130 Administered: All matched control subjects who enrolled in the study and following macimorelin administration.
Arm/Group | Cases/AEZS-130 Administered | Control/AEZS-130 Administered
Number analyzed (Participants) | 50 | 48
ng/mL | 2.36 (5.69) | 17.71 (19.11)
Statistical Analysis 1: Comparison: Cases/AEZS-130 Administered vs Control/AEZS-130 Administered; Summary of ROC Analyses following macimorelin administration; Test type: Other; ROC AUC = 0.923, 99% CI 1-sided [lower limit 0.850]
Statistical Analysis 2: Comparison: Cases/AEZS-130 Administered vs Control/AEZS-130 Administered; ROC analysis on peak GH concentrations in response to macimorelin: GH cut point of 2.7 ng/mL; Test type: Other — Sensitivity; sensitivity (percent) = 82
Statistical Analysis 3: Comparison: Cases/AEZS-130 Administered vs Control/AEZS-130 Administered; ROC analysis on peak GH concentrations in response to macimorelin: GH cut point of 2.7 ng/mL; Test type: Other — Specificity; Specificity (percent) = 92
Statistical Analysis 4: Comparison: Cases/AEZS-130 Administered vs Control/AEZS-130 Administered; ROC analysis on peak GH concentrations in response to macimorelin: GH cut point of 2.7 ng/mL; Test type: Other — Misclassification; misclassification (percent) = 13

2. Secondary Outcome: Peak Insulin-Like Growth Factor (IGF)-1 Concentration Following Treatment
Description: Descriptive summaries for IGF-1 and correlation with GH concentrations based on macimorelin treatment. Mean IGF-1 values taken pre- and post- macimorelin administration.
Time Frame: 15 min. before macimorelin administration and at 150 min after macimorelin administration
Population: Modified Intent-to-treat analysis set used for analysis of mean IGF-1 values taken pre- and post-macimorelin administration.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Case/AEZS-130 Administered: All AGHD patients who received macimorelin.
- Control/AEZS-130 Administered: All matched control subjects who received macimorelin.
Arm/Group | Case/AEZS-130 Administered | Control/AEZS-130 Administered
Number analyzed (Participants) | 52 | 48
ng/mL
  15 min before AEZS-130 | 58.1 (37.29) | 128.1 (52.47)
  150 min after AEZS-130 | 53.0 (34.57) | 125.9 (54.26)
Statistical Analysis 1: Comparison: Case/AEZS-130 Administered; Summary of IGF-1 before and after AEZS-130 administration: post - pre differences; Test type: Other; Mean Difference (Final Values) = -5.1, Standard Deviation 9.57
Statistical Analysis 2: Comparison: Control/AEZS-130 Administered; Test type: Other; Mean Difference (Final Values) = -2.3, Standard Deviation 16.25

3. Secondary Outcome: Classification and Regression Tree (CART) Analysis of Peak Growth Hormone (GH) Following Macimorelin Administration
Description: The CART Analysis for macimorelin estimated: a) a macimorelin cut-point that minimized the misclassification of AGHD patients and healthy control subjects; b) an optimal decision tree for macimorelin that incorporated age, sex and BMI.
  Sensitivity (correct identification of AGHD cases) and specificity (correct identification of control subjects) for macimorelin was summarized for age, gender, BMI and estrogen status subgroups containing n > 10.
  At least 8 of the 10 newly enrolled AGHD patients should have been correctly classified for a protocol pre-specified threshold of Peak GH concentration which was 8.5 (ng/ml).
  Software CART Version 6.0 was used.
Time Frame: GH sampling: pre-dose and 30, 45, 60, 75, 90, 120, 150 min post-dose
Population: PPS = per protocol set. Decision tree for sex abandoned. Following Amendment No. 4, no comparison with L-ARG + GHRH was performed.
Measure: Number; unit: percentage of participants
Groups:
- Peak GH: CART analysis of Peak GH following macimorelin administration
  Case Definition: GH ≤ 2.85 Control Definition: GH > 2.85
- Peak GH & BMI: CART analysis of Peak GH following macimorelin & BMI
  Case Definition: GH ≤ 2.85 or (2.85 <GH ≤7.15 & BMI ≤37.28) Control Definition: GH >7.15 or (2.85<GH≤7.15 and BMI>37.28)
- Peak GH & Age: CART analysis of Peak GH following macimorelin & Age
  Case Definition: GH ≤ 2.85 or (2.85 <GH ≤7.15 & age ≤47.5) Control Definition: GH > 7.15 or (2.85 <GH ≤7.15 & age >47.5)
- Peak GH & BMI & Age: CART analysis of Peak GH following macimorelin & BMI & Age
  Case Definition:
  GH≤0.85 or (0.85<GH≤2.85 and BMI>27.94) or (2.85<GH≤7.15 and age ≤47.5)
  Control Definition:
  GH > 7.15 or (0.85 <GH ≤2.85 & BMI ≤27.94) or (2.85<GH≤7.15 and age >47.5)
Arm/Group | Peak GH | Peak GH & BMI | Peak GH & Age | Peak GH & BMI & Age
Number analyzed (Participants) | 98 | 98 | 98 | 98
percentage of participants
  Misclassification | 13.3 | 11.2 | 10.2 | 9.2
  Sensitivity | 82.0 | 92.0 | 90.0 | 86.0
  Specificity | 91.7 | 85.4 | 89.6 | 95.8

4. Secondary Outcome: Number of Participants With Drug Related Adverse Events (AEs)
Description: Total number of participants with drug related AEs, following macimorelin administration of L-Arginine (ARG) - Growth Hormone Releasing Hormone (GHRH) administration.
Time Frame: 14 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- AGHD Patients (=Cases): All AGHD patients who were enrolled in this study.
- Match Control (= Control): All matched control subjects who were enrolled in the study.
Arm/Group | AGHD Patients (=Cases) | Match Control (= Control)
Number analyzed (Participants) | 53 | 48
Participants
  following AEZS-130 administration | 10 | 6
  following L-ARG+GHRH administration: number analyzed (Participants) | 43 | 10
  following L-ARG+GHRH administration | 19 | 3

ADVERSE EVENTS:
Time Frame: 14 days (time window between test visit (V2) and end-of-trial visit (V3)
Description: Only adverse events that occurred after the first dose of study drug (referred to as treatment-emergent adverse events (TEAEs)) were considered in the safety analysis. All treatment-emergent adverse events were summarized in terms of number and percentage of subjects and number and percentage of events within each treatment period by MedDRA system organ class and preferred term. A TEAE was attributed to the treatment that the subject received prior to the adverse event.
Groups:
- AEZS-130: Cases: All AGHD patients (cases) who received AEZS-130 (macimorelin).
- AEZS-130: Controls: All matched control subjects who received AEZS-130 (macimorelin).
- L-ARG+GHRH: Cases: All AGHD patients (cases) who received L-ARG+GHRH.
- L-ARG+GHRH: Controls: All matched control subjects who received L-ARG+GHRH.
Arm/Group | AEZS-130: Cases | AEZS-130: Controls | L-ARG+GHRH: Cases | L-ARG+GHRH: Controls
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/48 | 0/43 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/52 | 1/48 | 0/43 | 0/10
Other Adverse Events (participants affected / at risk) | 19/52 | 10/48 | 26/43 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AEZS-130: Cases (N=52) | AEZS-130: Controls (N=48) | L-ARG+GHRH: Cases (N=43) | L-ARG+GHRH: Controls (N=10)
ECG QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ECG T wave abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AEZS-130: Cases (N=52) | AEZS-130: Controls (N=48) | L-ARG+GHRH: Cases (N=43) | L-ARG+GHRH: Controls (N=10)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 10 (10) | 2 (2) | 6 (6) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ECG QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ECG T wave abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ECG change (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 16 (16) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomach discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinits (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Injection site irritation (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study Protocol Section 10.7 Draft versions of abstracts or manuscripts must be made available to the co-authors and to the sponsor before any presentation of results or submission for publication. At least 2 weeks should be allowed for review and comment of an abstract and 4 weeks in the case of a full paper, respectively.

Multiple review cycles are usual for full papers and respective planning must account for this.